CLINICAL TRIAL: NCT04696055
Title: An Open-Label Study of Regorafenib in Combination With Pembrolizumab in Patients With Advanced or Metastatic Hepatocellular Carcinoma (HCC) After PD1/PD-L1 Immune Checkpoint Inhibitors
Brief Title: Regorafenib Plus Pembrolizumab in Patients With Advanced or Spreading Liver Cancer Who Have Been Previously Treated With PD-1/PD-L1 Immune Checkpoint Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21469; MK-3475-B70 (Other: Merck); Keynote B70 (Other: Merck); 2020-003555-16 (EudraCT Number)
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2023-05-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Advanced or metastatic hepatocellular carcinoma (HCC); Liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — pembrolizumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib+Pembrolizumab (Experimental): Participants with advanced hepatocellular carcinoma (HCC) progressed on 1L anti-PD-1/PD-L1 therapy.
  Interventions: Drug: Pembrolizumab; Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 400 mg to be administered as an intravenous (IV) infusion every 6 weeks (Q6W).
  Other Names: Keytruda / MK-3475
Drug: Regorafenib (Stivarga, BAY73-4506) — Regorafenib to be given orally (p.o.) at a starting dose of 90 mg QD for 3 weeks of every 4 weeks (i.e., 3 weeks on, 1 week off). If the starting dose of 90 mg daily is well tolerated the dose should be escalated to 120 mg starting after the first 4-week cycle of regorafenib.

SUMMARY:
Researchers are looking for a better way to treat people diagnosed with liver cancer which may have spread to nearby tissue and is unlikely to be cured or controlled with treatment (advanced metastatic hepatocellular carcinoma, HCC). Before a treatment can be approved for people to take, researchers do clinical trials to better understand its safety and how it works.

In this trial, the researchers will learn more about the trial treatment, regorafenib, in a small number of participants. They will study the results when the trial treatment is taken with another cancer treatment called pembrolizumab.

There will be 2 parts to this trial. The part 1 (pilot phase) will include about 52 men and women. The part 2 (expansion phase) will include about 67 men and women. All of the participants will have HCC and will be aged 18 years or older. All of the participants will have tried other treatments that did not help their HCC. These other treatments (PD-1/PD-L1 Immune Checkpoint Inhibitors) are designed to work by stopping the activity of certain proteins in the immune system thought to play a role in HCC.

During both parts of the trial, the participants will take regorafenib and receive pembrolizumab. In the pilot phase, there will be 2 groups of participants. The group that each participant joins will be based on the treatment they already received for their HCC. The researchers will review the results in each group to learn if regorafenib and pembrolizumab are helping one group of participants more than others. Outcome of this review will determine the population to be treated in the expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age on the day of signing informed consent.
* Histological or cytological confirmation of HCC or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic participants.
* Unresectable advanced HCC eligible for systemic therapy.
* Participants must have progressed after only one prior line of systemic immunotherapy treatment with an anti-PD-1/PD-L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. A wash out period of at least 28 days or 5 half-lives, whichever is shorter, must be completed for eligibility in this trial. PD-1/PD-L1 treatment progression is defined by meeting all of the following criteria:

  1. Has received at least 2 doses of an approved anti PD-1/PD-L1 mAb or received PD-1/PD-L1 treatment for 8 weeks, whichever is longer.
  2. Has demonstrated disease progression after PD-1/PD-L1 treatment as defined by RECIST 1.1. In the absence of rapid clinical progression, the initial evidence of RECIST 1.1 disease progression is to be confirmed using iRECIST by a second assessment no less than four weeks from the date of the first documented progressive disease.

  i. This determination is made by the investigator. Once progressive disease is confirmed, the initial date of RECIST 1.1 progressive disease documentation will be considered that date of disease progression.

ii. In cases of unequivocal clinical or radiological progression, disease progression confirmation may not be required after documented discussion and approval by the sponsor.

c. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/PD-L1 mAb.

- Participants who receive anti-PD-1 therapy as adjuvant treatment following complete resection of liver cancer and have disease recurrence (unresectable locoregional disease or distant metastases) are eligible if they progressed while on active treatment or within 6 months of stopping anti-PD-1 therapy. This will be considered the first line of systemic therapy.

For these participants, the following applies:

1. a second assessment to confirm disease progression beyond recurrence is not required; and
2. they must have received at least 2 prior doses of anti-PD-1/PD-L1 mAb.

   * Barcelona Clinic Liver Cancer (BCLC) stage B or C.
   * Liver function status should be Child-Pugh (CP) Class A within 7 days prior to the first dose of study intervention. CP status should be calculated based on clinical findings and laboratory results during the screening period.
   * Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1 within 7 days prior to the first dose of study intervention.
   * At least one measurable lesion by CT scan or MRI according to RECIST 1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if there has been demonstrated progression in the lesion.
   * Participants with controlled (treated) hepatitis B virus (HBV) infection will be allowed if they meet the following criteria:

     * Antiviral therapy for HBV must be given for at least 4 weeks and HBV viral load must be less than 500 IU/mL prior to first dose of study intervention.
     * Participants on active HBV therapy with viral loads under 500 IU/ml should stay on the same therapy throughout study treatment.
     * Participants who are anti-HBc (+), negative for HBsAg, negative for anti-HBs, and have an HBV viral load under 500 IU/mL that do not require HBV antiviral prophylaxis.
   * Provision of recent tumor tissue (as defined below) is mandatory at screening. Exceptions will be accepted for participants with no recent baseline tumor tissues after documented discussion and approval by the sponsor.

     * Tumor tissue obtained within 180 days of enrollment and after the last dose of most recent anti-cancer therapy.
     * Or a new biopsy.

Exclusion Criteria:

* Fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes.
* Patients with disease that is suitable for local therapy administered with curative intent.
* Patients who experienced any Common Terminology Criteria for Adverse Events (CTCAE) ≥ 3 or any other immune- related toxicities that led to permanent discontinuation of treatment with immune checkpoint inhibitors in 1 L.
* Persistent proteinuria of CTCAE Grade 3 or higher.
* Diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study interventions.
* Active autoimmune disease.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Any hemorrhage or bleeding event CTCAE Grade ≥ 3 within 28 days prior to the start of study medication.
* Patients with large esophageal varices at risk of bleeding that are not being treated with conventional medical intervention.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication.
* Ongoing infection CTCAE Grade > 2 requiring systemic therapy.
* Dual active HBV infection (HBsAg (+) and / or detectable HBV DNA) and HCV infection (anti-HCV Ab (+) and detectable HCV RNA) at study entry.
* Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg) on more than 2 separate measurements despite optimal medical management.
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months).
* Myocardial infarction less than 6 months before start of study intervention.
* Pleural effusion or ascites that causes respiratory compromise (CTCAE Grade ≥ 2 dyspnea).
* Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 3 years prior to study entry.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable.
* Significant acute gastrointestinal disorders with diarrhea as a major symptom.
* Prior monotherapy treatment with any tyrosine kinase inhibitor in 1L.
* Prior treatment with regorafenib, in combination regimens with immune checkpoint inhibitors.
* Transfusion of blood products within 7 days prior to signing informed consent, or administration of colony stimulating factors within 4 weeks prior to signing informed consent.
* Previous assignment to treatment during this study.
* Previous (at least a minimum of 28 days, or 5 half-lives of an investigational drug before the start of study treatment, whichever is shorter) or concomitant participation in another clinical study with investigational medicinal product(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (9):
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope - Duarte Cancer Center, Duarte, California
  - USC Norris Hospital and Clinics, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - University of Miami Miller School of Medicine, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Seattle Cancer Care Alliance, Seattle, Washington
- France (9):
  - Hôpital Beaujon - Clichy, Clichy
  - Center Hospitalier Michallon - Grenoble, Grenoble
  - Hopital Claude Huriez - Lille, Lille
  - Hôpital de la Croix Rousse, Lyon
  - AP-HM - Hopital de la Timone, Marseille
  - Hôpital Saint-Eloi, Montpellier
  - Centre François Magendie - Pessac, Pessac
  - Centre Hospitalier Universitaire de Nancy, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse - Villejuif, Villejuif
- Germany (5):
  - Eberhard-Karls-Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München Grosshadern, München, Bavaria
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
- Israel (3):
  - Rambam Health Corporation, Haifa
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Humanitas Mirasole S.p.A., Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana_Santa Chiara - UO Oncologia 2, Pisa, Tuscany
  - Istituto Oncologico Veneto_Padova - UOC Oncologia 1, Padua, Veneto
- Japan (3):
  - Chiba University Hospital, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Japanese Red Cross Society Musashino Red Cross Hospital, Musashino, Tokyo
- South Korea (3):
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul
- Spain (3):
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón | Digestivo, Madrid

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/21469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 03 February 2021 (first participant first visit) and 23 April 2024 (last participant last visit) at 39 centers in 8 countries.
Pre-assignment Details: A total of 136 participants were screened, of whom 41 were screening failures. A total of 95 participants were assigned to treatment.
Groups:
- Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]): Cohort 1 with participants after one systemic line of therapy consisting of atezolizumab plus bevacizumab treatment combination only.
  Pembrolizumab 400 mg was administered as an intravenous (IV) infusion every 6 weeks. Regorafenib was given orally at a starting dose of 90 mg once daily for 3 weeks of every 4 weeks (i.e., 3 weeks on, 1 week off). If the starting dose of 90 mg daily was well tolerated the dose was escalated to 120 mg starting after the first 4-week cycle of regorafenib.
- Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment]): Cohort 2 with participants after one systemic line of therapy consisting of any PD-1/PD-L1 immune oncology (IO) containing first line treatment (excluding atezolizumab with or without bevacizumab) in monotherapy or combination regimens.
  Pembrolizumab 400 mg was administered as an IV infusion every 6 weeks. Regorafenib was given orally at a starting dose of 90 mg once daily for 3 weeks of every 4 weeks (i.e., 3 weeks on, 1 week off). If the starting dose of 90 mg daily was well tolerated the dose was escalated to 120 mg starting after the first 4-week cycle of regorafenib.
Period: Overall Study
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Started | 68 | 27
Completed | 0 | 0
Not Completed | 68 | 27
Not completed — Adverse Event | 10 | 2
Not completed — Death | 4 | 0
Not completed — Other | 7 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Progressive Disease - Clinical Progression | 1 | 1
Not completed — Progressive Disease - Radiological Progression | 42 | 20
Not completed — Subject Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who took at least 1 dose of study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment]) | Total
Number analyzed (Participants) | 68 | 27 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (13.1) | 70.9 (7.3) | 64.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 53 | 20 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 50 | 17 | 67
  Unknown or Not Reported | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 3 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 37 | 20 | 57
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per RECIST 1.1 by Central Assessment
Description: Overall response rate (ORR) is defined as the percentage of participants with best overall response of confirmed complete response (CR) or partial response (PR). ORR per RECIST 1.1 by independent central assessment is reported). RECIST 1.1: response evaluation criteria in solid tumors version 1.1
Time Frame: Up to 15 months. Data up to 38 months are now available and are also reported for full transparency.
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Number analyzed (Participants) | 68 | 27
Percentage of participants
  Up to 15 months (primary outcome as previously reported) | 5.9 [1.6 to 14.4] | 11.1 [2.4 to 29.2]
  Up to 38 months (as of study completion) | 7.4 [2.4 to 16.3] | 14.8 [4.2 to 33.7]

2. Secondary Outcome: Overall Response Rate (ORR) Per RECIST 1.1 by Investigator Assessment
Description: Overall response rate (ORR) is defined as the percentage of participants with best overall response of confirmed complete response (CR) or partial response (PR). ORR by RECIST 1.1 investigator review is reported. RECIST 1.1: response evaluation criteria in solid tumors version 1.1
Time Frame: Up to 38 months
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Number analyzed (Participants) | 68 | 27
Percentage of participants | 7.4 [2.4 to 16.3] | 18.5 [6.3 to 38.1]

3. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by Central Assessment and Investigator Assessment
Description: Duration of response (DOR) for partial response (PR) and complete response (CR) was defined as the time from the first documented objective response of PR or CR, whichever noted earlier, to disease progression or death (if death occurs before progression was documented). DOR was defined for confirmed responders only, i.e., participants with a CR or PR. RECIST 1.1: response evaluation criteria in solid tumors version 1.1
Time Frame: Up to 38 months
Population: Confirmed responders in Full Analysis Set (FAS)
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Number analyzed (Participants) | 5 | 5
Days
  Central assessment: number analyzed (Participants) | 5 | 4
  Central assessment | 210 [158 to 937] | 195 [83 to 280]
  Investigator assessment | 431 [82 to 893] | 364 [117 to 839]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was considered as treatment-emergent (TEAE) if arising or worsening after start of first study intervention administration until 30 days after administration of any study intervention. In addition, any AEs qualifying as a serious adverse event (SAE) were collected for 90 days after the last dose of pembrolizumab, unless a new anti-cancer therapy had been initiated.
Time Frame: Up to 38 months
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Number analyzed (Participants) | 68 | 27
Participants
  Any TEAE | 68 | 27
  Any SAE | 37 | 11

5. Secondary Outcome: Number of Participants With Safety-relevant Changes in Clinical Parameters
Description: Number of participants with clinically relevant trends observed in laboratory data, ECG data, or ECOG performance status is reported.
Time Frame: Up to 38 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Number analyzed (Participants) | 68 | 27
Participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Dose Modification
Description: Dose modification included dose interruption, dose reduction, dose discontinuation.
Time Frame: Up to 38 months
Population: Full Analysis Set (FAS)
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (Regorafenib + Pembrolizumab [1L: Atezolizumab + Bevacizumab]) | Cohort 2 (Regorafenib + Pembrolizumab [1L: Any Other IO Containing Treatment])
Number analyzed (Participants) | 68 | 27
Percentage of participants
  Regorafenib - drug interruptions or delays | 63.2 | 70.4
  Regorafenib - dose reductions | 41.2 | 63.0
  Regorafenib - drug withdrawal | 16.2 | 25.9
  Pembrolizumab - dose interruptions or delays | 14.7 | 25.9
  Pembrolizumab - drug withdrawal | 4.4 | 11.1

ADVERSE EVENTS:
Time Frame: These data extend to the final release date of the clinical database (38 months).
Description: All-Cause Mortality, Serious Adverse Events (SAEs) and Other Adverse Events were monitored from the start of study intervention until 30 days after the last administration of any study intervention. SAEs were additionally monitored for 90 days after last pembrolizumab infusion, unless a new anti-cancer therapy was initiated. All-Cause Mortality was also additionally monitored for 90 days after last pembrolizumab infusion.
Groups:
- Regorafenib+Pembrolizumab [1L: Atezolizumab + Bevacizumab]: Cohort 1 with participants after one systemic line of therapy consisting of atezolizumab plus bevacizumab treatment combination only. Pembrolizumab 400 mg was administered as an intravenous (IV) infusion every 6 weeks (Q6W). Regorafenib was given orally (p.o.) at a starting dose of 90 mg once daily (QD) for 3 weeks of every 4 weeks (i.e., 3 weeks on, 1 week off). If the starting dose of 90 mg daily was well tolerated the dose was escalated to 120 mg starting after the first 4-week cycle of regorafenib.
- Regorafenib+Pembrolizumab [Any Other IO Containing Treatment]: Cohort 2 with participants after one systemic line of therapy consisting of any PD-1/PD-L1 immune oncology (IO) containing first line treatment (excluding atezolizumab with or without bevacizumab) in monotherapy or combination regimens. Pembrolizumab 400 mg was administered as an intravenous (IV) infusion every 6 weeks (Q6W). Regorafenib was given orally (p.o.) at a starting dose of 90 mg once daily (QD) for 3 weeks of every 4 weeks (i.e., 3 weeks on, 1 week off). If the starting dose of 90 mg daily was well tolerated the dose was escalated to 120 mg starting after the first 4-week cycle of regorafenib.
Arm/Group | Regorafenib+Pembrolizumab [1L: Atezolizumab + Bevacizumab] | Regorafenib+Pembrolizumab [Any Other IO Containing Treatment]
All-Cause Mortality (participants affected / at risk) | 53/68 | 20/27
Serious Adverse Events (participants affected / at risk) | 37/68 | 11/27
Other Adverse Events (participants affected / at risk) | 63/68 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib+Pembrolizumab [1L: Atezolizumab + Bevacizumab] (N=68) | Regorafenib+Pembrolizumab [Any Other IO Containing Treatment] (N=27)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (3)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (5) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 2 (5)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (3) | 0 (0)
Meningorrhagia (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib+Pembrolizumab [1L: Atezolizumab + Bevacizumab] (N=68) | Regorafenib+Pembrolizumab [Any Other IO Containing Treatment] (N=27)
Anaemia (Blood and lymphatic system disorders) | 11 (22) | 2 (12)
Hypothyroidism (Endocrine disorders) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (17) | 5 (9)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 4 (6)
Ascites (Gastrointestinal disorders) | 5 (9) | 3 (3)
Constipation (Gastrointestinal disorders) | 14 (17) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 23 (37) | 13 (34)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (15) | 5 (8)
Stomatitis (Gastrointestinal disorders) | 5 (9) | 1 (3)
Vomiting (Gastrointestinal disorders) | 9 (10) | 3 (4)
Asthenia (General disorders) | 23 (52) | 18 (54)
Fatigue (General disorders) | 14 (21) | 4 (6)
Mucosal inflammation (General disorders) | 9 (9) | 4 (6)
Oedema peripheral (General disorders) | 8 (9) | 1 (1)
Pyrexia (General disorders) | 13 (16) | 5 (9)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (7) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 6 (7)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 9 (16) | 3 (7)
Blood bilirubin increased (Investigations) | 9 (13) | 6 (23)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 2 (3)
Lipase increased (Investigations) | 3 (7) | 2 (2)
Weight decreased (Investigations) | 7 (8) | 4 (8)
Transaminases increased (Investigations) | 4 (4) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (8) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (19) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (13) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 21 (32) | 13 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 10 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (12) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 5 (6) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (7) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 27 (64) | 14 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 10 (16) | 6 (12)
Hypertension (Vascular disorders) | 15 (23) | 9 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04696055/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04696055/SAP_002.pdf